PRIMROSE Trial – Informed Consent Form Version: 1.2

Study Code: IRAS number: **341315** Participant identification number:

Cardiothoracic Research Team,

Date: 17/03/25

Morriston Hospital, Swansea.

Principle Investigator: Tracy Jones



Study Title: A pilot study of a randomised controlled trial to evaluate the impact of thoracic PRehabilitation with Inspiratory Muscle TRaining Or Standard PrEhabilitation for surgical lung cancer patients. The PRIMROSE Trial

## **Informed Consent Form:**

Name of researcher: If you agree, please initial all the below boxes:

| I confirm that I have read the participant information sheet dated |
|---|
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected |
| I understand I can stop being part of the study at any time, without giving a reason, but information that we already have will be kept and used in the study. I understand no further information would be collected or any other research carried out |
| I understand that as part of the trial, initials/ NHS number/ name/ contact details including email address, will be collected so researchers can contact me and follow up on the research. I understand that individuals will use this information to do the research or to check records to make sure that the research is being done properly |
| I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from the Sponsor, Swansea Bay University Health Board where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records |
| As part of the trial, we will collect direct, anonymised quotations from participants. For example, how you managed with the device. I give permission for these anonymised quotations to be disseminated and published as part of the results of the study |
| I understand I will stop being part of the study if I lose capacity to provide ongoing consent and no further information will be collected. I give permission for collected information to be retained and used in the study |

<sup>\*1</sup>copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes.

| I agree to my General Practitioner being info | rmed of my participation i | n the study |
|---|---|---|
| I agree to take part in this study | | |
| Name of participant: | Date: | Signature: |
| Name of person taking consent: | Date: | Signature: |

Date: 17/03/25

Participant identification number:

PRIMROSE Trial – Informed Consent Form Version: 1.2

Study Code: IRAS number: **341315** 

<sup>\*1</sup>copy for participant; 1 copy for researcher site file; 1 (original) to be kept in medical notes.